CLINICAL TRIAL: NCT04620733
Title: RESPONSE: A Placebo-controlled, Randomized, Phase 3 Study to Evaluate the Efficacy and Safety of Seladelpar in Patients With Primary Biliary Cholangitis (PBC) and an Inadequate Response to or an Intolerance to Ursodeoxycholic Acid (UDCA)
Brief Title: RESPONSE: Response to Seladelpar in Subjects With Primary Biliary Cholangitis (PBC) and an Inadequate Control to or an Intolerance to Ursodeoxycholic Acid (UDCA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CB8025-32048; 2020-004348-27 (EudraCT Number)
Record Dates: First submitted 2020-11-04; First posted 2020-11-09 (Actual); Results first posted 2024-07-25 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Primary Biliary Cholangitis
Keywords: Primary Biliary Cholangitis (PBC); PBC
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — seladelpar

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive placebo to match seladelpar, orally, once daily, for a duration of up to 12 months.
  Interventions: Drug: Placebo
- Seladelpar (Experimental): Participants will receive seladelpar 10 mg (or 5 mg down-titrated, for those participants who met specific safety monitoring criteria or had tolerability issues), orally, once daily, for a duration of up to 12 months.
  Interventions: Drug: Seladelpar 10 mg; Drug: Seladelpar 5 mg

INTERVENTIONS:
Drug: Seladelpar 10 mg — Seladelpar 10 mg one capsule daily for double-blind period, for a duration of up to 12 months
  Arms: Seladelpar
Drug: Placebo — One capsule daily for double-blind period, for a duration of up to 12 months
  Arms: Placebo
Drug: Seladelpar 5 mg — If down-titration needed, one capsule daily for double-blind period, for a duration of up to 12 months
  Arms: Seladelpar

SUMMARY:
The purposes of this study are to evaluate the treatment effect of seladelpar on composite biochemical improvement in cholestasis markers based on ALP and total bilirubin and to evaluate the safety of seladelpar over 12 months of treatment compared to placebo.

The study also checked the effect of treatment on the symptoms of PBC, including pruritus.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have given written informed consent (signed and dated) and any authorizations required by local law.
* Male or female with a definitive diagnosis of primary biliary cholangitis (PBC).
* Ursodeoxycholic acid (UDCA) for the past 12 months (stable dose for >3 months prior to screening) or intolerant to UDCA (last dose of UDCA >3 months prior to screening).
* Laboratory parameters measured by the Central Laboratory at screening:

  * Alkaline phosphatase (ALP) ≥1.67× ULN (upper limit of normal)
  * Aspartate aminotransferase (AST) ≤3× ULN
  * Alanine aminotransferase (ALT) ≤3× ULN
  * Total bilirubin ≤2× ULN
  * Estimated glomerular filtration rate (eGFR) >45 mL/min/1.73 m^2 (calculated by the Modification of Diet in Renal Disease study equation).
  * International normalized ratio (INR) below 1.1× ULN (For individuals on anticoagulation therapy, INR must be maintained in the range required for prophylaxis for their specific disease).
  * Platelet count ≥100 ×10^3/µL.
* Females of reproductive potential must use at least 1 barrier contraceptive and a second effective birth control method during the study and for at least 90 days after the last dose. Male individuals who are sexually active with female partners of reproductive potential must use barrier contraception, and their female partners must use a second effective birth control method during the study and for at least 90 days after the last dose.

Key Exclusion Criteria:

* Previous exposure to seladelpar (MBX-8025).
* A medical condition other than PBC that, in the investigator's opinion, would preclude full participation in the study (e.g., cancer) or confound its results (e.g., Paget's disease, any active infection).
* Advanced PBC as defined by the Rotterdam criteria (albumin below the lower limit of normal and total bilirubin above 1.0 × ULN).
* Presence of clinically important hepatic decompensation, including the following:

  * History of liver transplantation, current placement on liver transplantation list, or current Model for End-Stage Liver Disease (MELD) score ≥12. For individuals on anticoagulation medication, evaluation of the baseline INR, in concert with their current dose adjustments of their anticoagulant medication, will be taken into account when calculating the MELD score. This will be done in consultation with the medical monitor.
  * Complications of portal hypertension, including known esophageal varices, history of variceal bleeds or related interventions (e.g., transjugular intrahepatic portosystemic shunt placement), ascites, and hepatic encephalopathy.
  * Cirrhosis with complications, including history or presence of spontaneous bacterial peritonitis, hepatocellular carcinoma, or hepatorenal syndrome.
* Other chronic liver diseases:

  * Current features of autoimmune hepatitis (AIH) as determined by the investigator based on immunoserology, liver biochemistry, or historic confirmed liver histology.
  * PSC determined by the presence of diagnostic cholangiographic findings.
  * History or clinical evidence of alcoholic liver disease.
  * History or clinical evidence of alpha-1-antitrypsin deficiency.
  * History of biopsy confirmed nonalcoholic steatohepatitis (NASH).
  * History or evidence of Gilbert's syndrome with elevated total bilirubin.
  * History or evidence of hemochromatosis.
  * Hepatitis B, defined as the presence of hepatitis B surface antigen.
  * Hepatitis C, defined as the presence of hepatitis C virus ribonucleic acid.
  * History, evidence, or high suspicion of hepatobiliary malignancy based on imaging, screening laboratory values, and/or clinical symptoms.
* Known history of human immunodeficiency virus (HIV) or positive antibody test at screening
* Clinically important alcohol consumption, defined as more than 2 drink units per day (equivalent to 20 g) in women and 3 drink units per day (equivalent to 30 g) in men, or inability to quantify alcohol intake reliably.
* History of malignancy diagnosed or treated, actively or within 2 years, or ongoing evaluation for malignancy; localized treatment of squamous or noninvasive basal cell skin cancers and cervical carcinoma in situ is allowed if appropriately treated prior to screening.
* Treatment with obeticholic acid (OCA) or fibrates (e.g., bezafibrate, fenofibrate, elafibranor, lanifibranor, pemafibrate, saroglitizar) 6 weeks prior to screening.
* Treatment with colchicine, methotrexate, azathioprine, or long-term systemic corticosteroids (>2 weeks) during 2 months prior to screening
* Treatment with anti-pruritic drugs (e.g., cholestyramine, naltrexone, rifampicin, sertraline, or any experimental approach) must be on a stable dose within 1 month prior to screening
* Treatment with any other investigational therapy or device within 30 days or within 5 half-lives, whichever is longer, prior to screening
* For females, pregnancy or breastfeeding.
* Any other condition(s) that would compromise the safety of the individual or compromise the quality of the clinical study, as judged by the investigator.
* Immunosuppressant therapies.
* Other medications that effect liver or gastrointestinal (GI) functions, such as absorption of medications or the roux-en-y gastric bypass procedure, may be prohibited and should be discussed with the medical monitor on a case-by-case basis.
* Active Coronavirus Disease-2019 (COVID-19) infection during Screening.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CymaBay Study Director, Study Director — Gilead Sciences
Locations (134):
- United States (40):
  - The Institute for Liver Health DBA Arizona Liver Health, Chandler, Arizona
  - Arkansas Diagnostic Center, Little Rock, Arkansas
  - Stanford University School of Medicine, Palo Alto, California
  - California Liver Research Institute, Pasadena, California
  - University of California, Davis Medical Center, Sacramento, California
  - California Pacific Medical Center - Sutter Pacific Medical Foundation, San Francisco, California
  - Covenant Metabolic Specialists, LLC, Fort Myers, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - Covenant Research and Clinics, LLC, Sarasota, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Hospitals, Chicago, Illinois
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Novi, Michigan
  - MNGI Digestive Health, P.A., Maplewood, Minnesota
  - Southern Therapy and Advanced Research, LLC (STAR), Jackson, Mississippi
  - Saint Louis University, St Louis, Missouri
  - NYU Langone Health / NYU Grossman School of Medicine, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Care Access Research - Lumberton, Lumberton, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC Center for Liver Diseases, Pittsburgh, Pennsylvania
  - Galen Hepatology, Chattanooga, Tennessee
  - Gastro One, Germantown, Tennessee
  - Vanderbilt Digestive Disease Center, Nashville, Tennessee
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Digestive Disease Consultants dba GI Alliance, Fort Hood, Texas
  - Baylor College of Medicine, Houston, Texas
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
  - Pinnacle Clinical Research, PLLC, San Antonio, Texas
  - Bon Secours Richmond Community Hospital LLC, Richmond, Virginia
  - Liver Institute Northwest, Seattle, Washington
- Argentina (6):
  - Centro Medico Dra. De Salvo, CABA, Buenos Aires
  - STAT Research S.A., Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - DIM CliniaPrivada, Ramos Mejía, Buenos Aires
  - CINME (Centro de Investigaciones Metabolicas), Buenos Aires
  - Hospital Italiano de Buenos Aires, Caba
- Australia (4):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Klinikum Wels-Grieskirchen GmbH, Abteilung Fur Innere Medizin I - Gastroenterologie, Wels, Austria
- Belgium (5):
  - UZ Antwerpen, Edegem, Antwerpen
  - CHU de Liège, Liège, Liège
  - AZ Maria Middelares, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - Universitaire Ziekenhuizen Leuven, Leuven, Vlaams-Brabant
- Canada (3):
  - London Health Sciences Centre, London, Ontario
  - University Health Network, Toronto, Ontario
  - Toronto Digestive Disease Associates Inc, Vaughan, Ontario
- Chile (3):
  - Centro Clinico Mediterraneo, La Serena, Coquimbo Region
  - Clinical Research Chile SpA, Valdivia, Los Ríos Region
  - Centro de Investigaciones Clínicas Vina del Mar, Valparaíso
- Fakultni nemocnice Ostrava- Interni a Kardiologicka Klinika, Oddeleni gastroenterologie, hepatologie a pankreatologie, Ostrava, Czechia
- Denmark (2):
  - Aalborg Universitetshospital, Ambulatoriet for Medicinske Mave-Tarm Sygdomme, Aalborg
  - Hvidovre Hospital, Hvidovre
- France (3):
  - CHU de Grenoble, Grenoble
  - Hopital de la Croix-Rousse, Lyon
  - Hopital Saint-Antoine - Service d'Hepato-Gastro-Enterologie -184, rue du Faubourg Saint-Antoine, Paris
- Germany (7):
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum des Saarlandes, Homburg, Saarland
  - Universitatsklinikum Erlangen, Medizinische Klinik I, Gastroenterologie, Erlangen
  - Universitatsklinikum Frankfurt. Medizinische Klinik I, Frankfurt am Main
  - Ifi-Medizin GmbH, Hamburg
  - Gastroenterologische Gemeinschaftspraxis, Herne
  - Universitatsklinikum Leipzig, Leipzig
- Greece (2):
  - Ippokrateio General Hospital of Athens, Athens, Attica
  - General University Hospital of Larissa Department of Medicine and Research Laboratory of internal rv1edicine, National Expertise Center of Greece in Autoimmune liver Diseases, Larissa
- Hungary (2):
  - Semmelweis Egyetem, Budapest
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
- Israel (3):
  - Liver Unit, Jerusalem
  - Liver Disease Center, Sheba Medical Center, Ramat Gan
  - Institute for Digestive Tract & Liver Disease, Tel Aviv
- Italy (6):
  - ASST di Monza, Monza, MB
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona-Umberto I G.M. Lancisi G. Salesi, Ancona
  - Nuovo Ospedale Civile S. Agostino-Estense di Baggiovara, Bologna
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Azienda Ospedaliera Universita Padova, Padua
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
- Mexico (4):
  - Consultorio de la Doctora Maria Sarai Gonzalez Huezo, Metepec
  - Campeche No. 280, Int. 601 y 602, Col. Hipodromo, Cuauhtemoc, Mexico City
  - Consultorio Medico - Distrito Federal, Mexico City
  - Hospital Universitario Dr. Jose Eleuterio González, Monterrey
- New Zealand (2):
  - Gastroenterology, Christchurch Hospital, Christchurch, Canterbury
  - Gastroenterology Research Unit Dunedin Hospital, Dunedin, Otago
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne Im., Katowice
  - ID Clinic Akradiusz Pisula, Mysłowice
- Fundeni Clinical Institute, Bucharest, Romania
- Russia (6):
  - State budget institution of healthcare of Moscow city "Moscow Clinical Scientific and Practical Centre n. a. A.S. Loginov" of Moscow City Healthcare, Department, Central Research Institute of Gastroenterology, Moscow
  - Federal State Autonomous Educational Institution of Higher Education "Peoples' Friendship University of Russia", Centre of Liver Studies, Moscow
  - Clinic of High Medical Technologies n.a. N.I. Pirogov, Saint Petersburg
  - LLC Medical Company "Hepatolog", Samara
  - Stavropol state medical university, Stavropol
  - Ulyanovsk Regional Clinical Hospital, Ulyanovsk
- South Korea (9):
  - Inje University Busan Paik Hospital, Busan, Busan Gwangyeogsi
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si, Gyeonggido
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital Yonsei University Health System - PPDS, Soeul
- Spain (6):
  - Hospital Universitario German Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Margues de Valdecilla, Santander, Cantabria
  - Hospital Universitario Virgen de la Victoria, Málaga, Malaga
  - Hospital Universitario Vall D'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- University of Zurich, Gastroenterology and Hepatology, Zurich, Switzerland
- Turkey (Türkiye) (5):
  - Ankara Gazi University Faculty of Medicine Hospital, Ankara
  - Ankara Sehir Hastanesi, Ankara
  - Bezmi Alem University, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - Ege University Medical Faculty, Izmir
- Ukraine (2):
  - Municipal Non-profit Enterprise "City Clinical Hospital #13" of Kharkiv City Council, Kharkiv
  - Medical Center OK!Clinic+LLC International Institute of Clinical Research, Kyiv
- United Kingdom (8):
  - University Hospitals Plymouth NHS Trust, Plymouth, Devon
  - Portsmouth Hospitals NHS Trust, Portsmouth, Hampshire
  - Barts Health NHS Trust, Royal London Hospital, Ambrose King Centre, London, London, City of
  - Queen's Medical Centre, Nottingham, Nottinghamshire
  - Gemini Clinical Trial Unit, Oxford, Oxfordshire
  - University Hospitals Birmingham NHS Foundation Trust, Heritage Building (Queen Elizabeth Hospital), Birmingham
  - Hull Royal Infirmary, Hull
  - Kings College Hospital, London

REFERENCES:
- [Derived] Hirschfield GM, Bowlus CL, Mayo MJ, Kremer AE, Vierling JM, Kowdley KV, Levy C, Villamil A, Ladron de Guevara Cetina AL, Janczewska E, Zigmond E, Jeong SH, Yilmaz Y, Kallis Y, Corpechot C, Buggisch P, Invernizzi P, Londono Hurtado MC, Bergheanu S, Yang K, Choi YJ, Crittenden DB, McWherter CA; RESPONSE Study Group. A Phase 3 Trial of Seladelpar in Primary Biliary Cholangitis. N Engl J Med. 2024 Feb 29;390(9):783-794. doi: 10.1056/NEJMoa2312100. Epub 2024 Feb 21. PMID 38381664

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the Asia Pacific, Europe, Latin America, and North America.
Pre-assignment Details: 360 participants were screened.
Groups:
- Placebo: Participants received placebo to match seladelpar, orally, once daily, for a duration of up to 12 months.
- Seladelpar: Participants received seladelpar 10 mg, orally, once daily, for a duration of up to 12 months.
Period: Overall Study
Arm/Group | Placebo | Seladelpar
Started | 65 | 128
Completed | 57 | 117
Not Completed | 8 | 11
Not completed — Adverse Event | 4 | 3
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Deviation | 1 | 1
Not completed — Reason Not Specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set was defined as any participant who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Seladelpar | Total
Number analyzed (Participants) | 65 | 128 | 193
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 99 | 152
  >=65 years | 12 | 29 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (9.2) | 57 (10.0) | 57 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 123 | 183
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 29 | 56
  Not Hispanic or Latino | 38 | 97 | 135
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 4 | 7 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 56 | 114 | 170
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 48 | 61
  Argentina | 13 | 16 | 29
  Mexico | 6 | 6 | 12
  Spain | 4 | 7 | 11
  Russia | 1 | 8 | 9
  Italy | 4 | 4 | 8
  Turkey | 1 | 7 | 8
  United Kingdom | 2 | 6 | 8
  Poland | 5 | 2 | 7
  South Korea | 3 | 4 | 7
  Israel | 2 | 3 | 5
  Belgium | 2 | 1 | 3
  Czechia | 1 | 2 | 3
  Switzerland | 2 | 1 | 3
  Australia | 1 | 1 | 2
  Canada | 0 | 2 | 2
  Chile | 0 | 2 | 2
  France | 0 | 2 | 2
  Germany | 1 | 1 | 2
  Greece | 2 | 0 | 2
  Hungary | 0 | 2 | 2
  New Zealand | 2 | 0 | 2
  Romania | 0 | 2 | 2
  Austria | 0 | 1 | 1
Pruritus Numerical Rating Scale (NRS) for Participants With Baseline Pruritus NRS ≥ 4 [Mean (Standard Deviation); unit: score on a scale] — Population: Moderate to Severe Pruritus NRS (MSPN) Analysis Set included participants in the Intent-to-Treat (ITT) Analysis Set who had a baseline NRS value.
  score on a scale
    number analyzed (Participants) | 23 | 49 | 72
    (all) | 6.6 (1.44) | 6.1 (1.42) | 6.3 (1.43)
Alkaline Phosphatase (ALP) Levels [Mean (Standard Deviation); unit: U/L] | 313.8 (117.68) | 314.6 (122.96) | 314.3 (120.90)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response Criteria for the Composite Endpoint of ALP <1.67 × Upper Limit of Normal (ULN), ≥15% Reduction in ALP, and Total Bilirubin ≤ 1.0× ULN at Month 12
Description: Percentages were rounded-off.
Time Frame: Month 12
Population: The Intend-to-treat Analysis Set was defined as any participant who was randomized into the study and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Seladelpar
Number analyzed (Participants) | 65 | 128
percentage of participants | 20.0 [10.3 to 29.7] | 61.7 [53.3 to 70.1]
Statistical Analysis 1: Comparison: Placebo vs Seladelpar; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Two-sided p-value for pair-wise comparison was based on the CMH test adjusted for both randomization stratification variables (baseline ALP level: < 350 U/L and ≥ 350 U/L; baseline Pruritus NRS: < 4 and ≥ 4); Risk Difference (RD) = 41.7, 95% CI 2-sided [27.7 to 53.4]

2. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: Percentages were rounded-off.
Time Frame: First dose date up to last dose plus 30 days (up to 13.4 months)
Population: The Safety Analysis Set was defined as any participant who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Seladelpar
Number analyzed (Participants) | 65 | 128
percentage of participants
  TEAEs | 84.6 | 86.7
  Serious TEAEs | 6.2 | 7.0

3. Primary Outcome: Percentage of Participants With Shift of ≥ 2 CTCAE Grades From Baseline in Treatment-emergent Laboratory Abnormalities Related to Hematology and Select Liver Biochemistry
Description: Treatment-emergent graded laboratory abnormalities were defined as values that increase at least 2 toxicity grade from baseline at any time post baseline. The laboratory abnormalities were graded using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), where Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: potentially life-threatening laboratory abnormality.
  The data is reported for shift of ≥ 2 grades from baseline in values for hematology and select liver biochemistry. Hematology includes parameters like RBCs, (erythrocytes), hemoglobin, hematocrit, platelets, WBC, WBC differentials (absolute and percentage) including basophils, neutrophils, lymphocytes, eosinophils, and monocytes, etc. Biochemistry included select liver function tests like blood bilirubin, gamma-glutamyl transferase (GGT), aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase. Percentages were rounded-off.
Time Frame: First dose date up to last dose (up to 13.4 months)
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Seladelpar
Number analyzed (Participants) | 65 | 128
percentage of participants
  Shift ≥ 2 CTCAE grades in haematology | 12.3 | 14.1
  Shift ≥ 2 CTCAE grades in biochemistry | 6.2 | 7.0

4. Secondary Outcome: Percentage of Participants With ALP ≤1.0× ULN at Month 12
Description: Percentages were rounded-off.
Time Frame: Month 12
Population: Participants in Intent-to-treat Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Seladelpar
Number analyzed (Participants) | 65 | 128
percentage of participants | 0.0 [0.0 to 0.0] | 25.0 [17.5 to 32.5]
Statistical Analysis 1: Comparison: Placebo vs Seladelpar; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 25.0, 95% CI 2-sided [18.3 to 33.2] — Two-sided p-value for pair-wise comparison is based on the Cochran Mantel Haenszel test adjusted for both stratification variables (baseline ALP level: < 350 U/L and >= 350 U/L; baseline pruritus NRS: < 4 and >= 4)

5. Secondary Outcome: Change From Baseline in Weekly Averaged Pruritus Numerical Rating Scale (NRS) in Participants With NRS ≥ 4 at Month 6
Description: Pruritus NRS is used to rate the intensity of the itching experienced by the participants in the past 24 hours from no itching to worst possible itching by selecting a number from 0 to 10 on Itch Scale. Zero means no itching and 10 means worst imaginable itching.
Time Frame: Baseline, Month 6
Population: The Moderate to Severe Pruritus NRS Analysis Set included participants in the Intent-to-treat Analysis Set who had a baseline NRS value ≥ 4. Participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Seladelpar
Number analyzed (Participants) | 20 | 45
score on scale | -1.7 (0.41) | -3.2 (0.28)
Statistical Analysis 1: Comparison: Placebo vs Seladelpar; Test type: Superiority; p = 0.0047, MMRM; Mixed-Effect Model Repeated Measure (MMRM); Least Squares (LS) Mean Difference = -1.5, 95% CI 2-sided [-2.5 to -0.5]

ADVERSE EVENTS:
Time Frame: All-cause mortality: Up to 20.6 months; Adverse events: Up to last dose plus 30 days (Up to 13.4 months)
Description: All-cause mortality: All-Randomized Analysis Set was defined all participants randomized in the study.
  Adverse events: The Safety Analysis Set was defined as any participant who received at least 1 dose of study drug.
  There was only 1 participant who was down-titrated to the 5 mg seladelpar dose during the study. Therefore, the data for adverse events at 5 mg dose were not reported due to participant's confidentiality reasons.
Arm/Group | Placebo | Seladelpar
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/128
Serious Adverse Events (participants affected / at risk) | 4/65 | 9/128
Other Adverse Events (participants affected / at risk) | 40/65 | 66/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=65) | Seladelpar (N=128)
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Covid-19 (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=65) | Seladelpar (N=128)
Vertigo positional (Ear and labyrinth disorders) | 4 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 8
Abdominal pain (Gastrointestinal disorders) | 1 | 9
Nausea (Gastrointestinal disorders) | 3 | 8
Asthenia (General disorders) | 4 | 5
Fatigue (General disorders) | 4 | 8
Covid-19 (Infections and infestations) | 9 | 23
Nasopharyngitis (Infections and infestations) | 5 | 7
Pharyngitis (Infections and infestations) | 5 | 4
Upper respiratory tract infection (Infections and infestations) | 6 | 1
Urinary tract infection (Infections and infestations) | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 8
Headache (Nervous system disorders) | 1 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 6
Hypertension (Vascular disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/33/NCT04620733/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/33/NCT04620733/SAP_001.pdf